CLINICAL TRIAL: NCT04233827
Title: Mobile Biosensor for Measuring Vital Signs in Healthcare and Home Settings
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sara H. Browne, MD, MPH, Professor, University of California, San Diego
Other Study IDs: 161573
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2022-12

CONDITIONS: Pulse Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will record vital signs (heart rate and blood oxygen levels) using a new cell phone integrated biosensor and compare it to routine measurements carried out in the clinics and hospital at UCSD. Cell phones will be given to a selected group of subjects for use at home and data collected.

DETAILED DESCRIPTION:
Maxim Vital Sign study is a 2 part, investigator initiated observational study with Maxim Integrated aimed to compare vital sign readings using 2 prototype versions of new cell phone based mobile biosensors with standard of care (SOC). Adult subjects will be recruited from UCSD outpatient clinics, AVRC clinic, emergency department (ED), and hospitals. Vital signs will be measured using cell phone based mobile biosensors and SOC.

For Phase 1, up to 800 subjects will be recruited (700 adults and up to 100 adolescents). 250 subjects (200 adults and up to 50 adolescents) will participate in phase 1a and 550 subjects (500 adults and up to 50 adolescents) will participate in phase 1b. An additional group of 30 adult subjects will be recruited from outpatient clinics for participation in phase 2.

Phase 1a:

Two identical copies of the device will be tested during the first part of phase 1 with a total of 125 subjects (100 adults and up to 25 adolescents). Each prototype version will be tested on up to 125 subjects (100 adults and 25 adolescents) and compared to readings obtained by Welch-Allyn Spot Vital Signs monitor. Data will be obtained on the usability and accuracy of the measurements with each initial prototype. Measurement particularly of SpO2 depends on accurate finger position. Current SpO2 monitors encase the finger and immobilize it in order to obtain an accurate measurement. Maxim Integrated, in collaboration with DD Studios, Carlsbad CA, and Specialists in Global Health, Encinitas CA, have developed prototypes, which will be tested to inform design flaws in future prototypes.

Phase 1b:

Based on the results from phase 1a, one of the prototypes will be selected for further testing (the one with the least within-instrument variation). During Phase 1b, vital sign readings will be collected with the selected Maxim biosensor prototype and one of the Welch-Allyn Spot Vital Signs monitor simultaneously. The subjects will be recruited from both outpatient and hospital settings for accuracy and usability. A total of 550 subjects (500 adults and 50 adolescents) will be recruited for this part of phase 1.

ELIGIBILITY:
Inclusion Criteria:

1. Children (≥ 13 years old) and adult male and female subjects who provide written informed consent and assent.
2. Subjects must be willing to use the mobile device and answer questions regarding their experience.

Exclusion Criteria:

Individuals with prior or recent injury to one or both of their index fingers that would prevent or interfere with the use of Maxim biosensor.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children (≥ 13 years old) and adult male and female subjects who provide written informed consent and assent.
Sampling Method: Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of vital signs (HR and SpO2) | 20 minutes
  The accuracy of the vital sign (HR and SpO2) readings collected by Maxim biosensor compared to standard of care Welch-Allyn Spot Vital Sign monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Sara H Browne, MD MPH, Principal Investigator — UC San Diego
Locations (1):
- UCSD AntiViral Research Center, San Diego, California, United States

REFERENCES:
- [Derived] Browne SH, Bernstein M, Pan SC, Gonzalez Garcia J, Easson CA, Huang CC, Vaida F. Smartphone Biosensor With App Meets FDA/ISO Standards for Clinical Pulse Oximetry and Can Be Reliably Used by a Wide Range of Patients. Chest. 2021 Feb;159(2):724-732. doi: 10.1016/j.chest.2020.08.2104. Epub 2020 Sep 11. PMID 32926871